CLINICAL TRIAL: NCT06261242
Title: A Study of Tripod-Fix Vertebral Body Augmentation System in Vertebral Compression Fractures Caused by Osteoporosis
Brief Title: Tripod-Fix Vertebral Body Augmentation System in Osteoporotic Vertebral Compression Fractures Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Cheng-Li Lin, Director of Spinal Division/Associate Professor, National Cheng-Kung University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TWM-C-2201
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-02

CONDITIONS: Osteoporotic Vertebral Compression Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Tripod-Fix will be used to treat osteoporotic vertebral compression fractures.
  Interventions: Device: Tripod-Fix Vertebral Body Augmentation System (Tripod-Fix)

INTERVENTIONS:
Device: Tripod-Fix Vertebral Body Augmentation System (Tripod-Fix) — The Tripod-Fix is a permanent implant used for vertebral augmentation in patients with osteoporotic vertebral compression fractures.

SUMMARY:
This study is to evaluate the safety and effectiveness of the Tripod-Fix with Tecres Mendec® Spine HV System to treat subjects with osteoporotic vertebral compression fractures.

DETAILED DESCRIPTION:
This study is a prospective, single-center, open-label, single-arm study. This study will screen up to 12 eligible patients. Eligible patients will be treated with Tripod-Fix on the Day 1 and follow-up for 12 months. Patients will be asked to return to the study site for assessments on the Day 5, 1st month, 6th month and 12th month. Safety will be assessed by the investigator(s) at each return visit and will be monitored until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form prior to any study procedures.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female with at least 50 years of age.
4. 1 painful VCF which meet all of the following criteria:

   1. Fracture due to diagnosed or presumed underlying osteoporosis (T-score < -2.5 points).
   2. VCF between T7 and L4.
   3. Fracture age < 3 months.
   4. VCF shows loss of height in the anterior, mid or posterior third of the vertebral body from an estimated pre-fracture configuration of at least 15% but not more than 40% based on X-ray, CT or MRI at baseline.
   5. The Index fracture is acute or persistent (not healed), as demonstrated by MRI or bone scan.
5. Patient has failed conservative medical therapy, complementary and alternative medicine, defined as either having a VAS back pain score of ≥ 50 mm at 6 weeks after initiation of fracture care or a VAS back pain score of ≥ 70 mm at 2 weeks after initiation of fracture care. If patients with pain ≥ 70 mm at baseline continued to deteriorate as demonstrated by increasing VAS score and/or progressive vertebral collapse, treatment might be initiated after 1 week of conservative care.
6. Investigator believes target vertebral body is suitable for Tripod-Fix procedure (e.g., appropriate pedicle diameter) assessed on radiography preoperative.
7. Patient has an ODI score of ≥ 30/100.

Exclusion Criteria:

1. Target VCF due to high-energy trauma or underlying/suspected tumor.
2. Target VCF is diagnosed as an osteonecrosis.
3. Segmental kyphosis of target vertebral compression > 30°.
4. Any prior surgical treatment for a VCF or other surgical procedure on the target vertebral body or adjacent level.
5. The patient has uncontrolled systemic diabetes (A1c > 10) and /or uncontrolled hypertension (patient requiring 3 or more anti-hypertensive drugs).
6. Pre-existing or clinically unstable neurologic deficit.
7. Spinal canal compromise causing clinical manifestations of cord, neural foramen, or nerve root compression at the level to be treated.
8. Any physical exam evidence of myelopathy, radiculopathy, or coagulopathy.
9. Disabling back pain due to causes other than acute fracture, or any other condition that requires daily narcotic medication, such as clinical diagnosis of herniated nucleus pulposus or severe spinal stenosis (progressive weakness or paralysis).
10. Patient not able to walk without assistance prior to fracture.
11. Any radiographic evidence of cortical disruption, burst fractures and pedicle fracture.
12. Translation > 4 mm or Spondylolisthesis > Grade 1 at target vertebral body.
13. Any underlying systemic bone disease other than osteoporosis (e.g., osteomalacia, osteogenesis imperfect, Paget's disease, etc.).
14. In the investigator's opinion, a patient with any other medical illness or condition which may not be suitable to participate in the study, including but not limited to: A medical contraindication to spinal surgery and/or general anesthesia, such as Patients on chronic anti-coagulation. (Patients stop the treatment 8 days before surgery with a threshold for normal being INR < 1.1 and platelets > 100,000 are not limited to this.)
15. Prior history of intolerance or allergic reaction to titanium and/or one of the components of the PMMA cement.
16. Active systemic or local infection at baseline.
17. Body mass index > 40.
18. Patients affected by severe cardiopulmonary deficiencies.
19. In the investigator's opinion, a patient with any other medical illness or condition which may not be suitable to participate in the study, including but not limited to: Likely to impair long-term follow-up (e.g., cancer).
20. Any evidence of alcohol or drug abuse.
21. Uncontrolled psychiatric disorders are defined by the DSM V or severe dementia.
22. Currently on anti-cancer therapy or anti-HIV therapy.
23. Life expectancy is less than the study duration or undergoing palliative care.
24. Participating in any other investigational study.
25. On long-term steroid therapy (steroid dose ≥ 30 mg /day for > 3 months).
26. Known to be involved in spinal litigation.
27. Pregnant women as confirmed by positive pregnancy test or considering getting pregnant during study participation.
28. Presenting loss of vertebral height > 50% compared to estimated pre-fracture height.
29. Interspinous-process widening.
30. Sclerotic fracture or pseudarthrosis.
31. Patient is a prisoner or not in the wards of the court.
32. Patients with contraindications to MRI and bone scan.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with study success | 12 months post-procedure
  To evaluate the safety and effectiveness of the Tripod-Fix with treatment success defined as a subject must meet all the components of primary composite endpoint:
  1. The reduction of Visual Analogue Scale (VAS) score > 20 mm at the 12th month from the Baseline as measured by the 100-mm VAS measurement, AND
  2. Maintenance or improvement in function at the 12th month from the Baseline as measured by the 100-point Oswestry Disability Index (ODI), AND
  3. Absence of device-related serious adverse events, defined as the following events with the evidence in radiological parameters: device-related adverse events (device migration, recollapse, protrusion), or symptomatic cement extravasation requiring surgical reintervention or retreatment at the index level, including revision, removal, reoperation, and/or supplemental fixation.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Li Lin, Principal Investigator — NCKUH Department of Orthopedics
Locations (1):
- National Cheng Kung University Hospital Department of Orthopedics, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No